CLINICAL TRIAL: NCT04314089
Title: Phase Ib First in Human Dose Escalation of GT103 in Refractory, Advanced Stage Non-Small Cell Lung Cancer (TOP 1902)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edward Patz (Other)
Responsible Party: Sponsor-Investigator, Edward Patz, James and Alice Chen Distinguished Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00104564
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Stage III/IV NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GT103 (Experimental): Participants will receive GT103 every 3 weeks. GT103 will be escalated from .3mg/kg up 10 to mg/kg or until MTD is found
  Interventions: Drug: GT103

INTERVENTIONS:
Drug: GT103 — intravenously (dose depending)

SUMMARY:
The purpose of this research study is to determine the maximum tolerated dose of GT103 and investigate the safety and effectiveness of the study drug.

DETAILED DESCRIPTION:
This is a Phase Ib First in Human Dose Escalation of GT103 in Refractory, Advanced Stage (III/IV) and Recurrent Non-Small Cell Lung Cancer.

Patients with histologically confirmed recurrent, advanced stage of lung cancer, and there are no other standard therapies available may be eligible to participate in this study.

ELIGIBILITY:
Inclusion Criteria;

1. Histologically and/or cytologically confirmed advanced stage III, IV or recurrent NSCLC whose tumors have progressed on prior therapy.
2. Prior Therapy:

   * Patients must have received immunotherapy (anti-PD-1/PD-Ll) and a platinum- based chemotherapy either concomitantly or sequentially. There is no defined window of time since receiving immunotherapy. Immunotherapy does not have to be the immediate treatment prior to this protocol therapy.
   * Patients with EGFR, ALK, or ROS1 alterations must have received at least one prior TKI and prior chemotherapy (at least one platinum doublet regimen).
   * Stage III patients:

   If previously treated with immunotherapy participants with investigator-assessed radiographic disease progression or recurrence in less than 6 months after the last dose of immunotherapy in Stage III B/C disease post concurrent chemoradiotherapy followed by immunotherapy are eligible. Radiographic progression must be documented via pretreatment scan as compared to the prior therapy baseline scan in order for the participant to be eligible.
3. Disease must be measurable by RECIST 1.1 criteria (see Appendix A). Tumor lesions in a previously irradiated area are considered measurable IF progression has been demonstrated in such lesions after radiation.
4. Age ≥ 18 years
5. ECOG Performance Status 0 or 1 (see Appendix B)
6. Adequate bone marrow function as shown by:

   * ANC ≥ 1.5 x 109
   * Platelets ≥ 100 x 109/L
   * Hemoglobin ≥ 9 g/dL; Erythropoietin and transfusion support is permitted. If patient is receiving supportive care, hemoglobin must be stable above or equal to 9 g/dL for at least 2 weeks prior to day 1 of study drug without blood transfusion to maintain hemoglobin level.
7. Adequate liver function as shown by:

   * serum bilirubin ≤ 1.5x ULN
   * ALT and AST ≤ 2.5x ULN ; ≤ 5 x ULN with liver metastasis
8. Adequate renal function: defined as creatinine clearance (estimated) ≥ 50 cc/min by Cockroft Gault or 24-hour urine (see Appendix E).
9. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and prior to treatment on Cycle 1 Day 1; both men and women must be willing to use two medically accepted methods of contraception, one of them being a barrier method during the study and for 6 months after last study drug administration. See Section 6.3.1.1 for a list of acceptable methods of contraception.
10. Signed informed consent
11. Willing and able to comply with clinic visits and study-related procedures and requirements.

Exclusion Criteria;

1. Patients currently receiving anticancer therapies or who have received anticancer therapies within 2 weeks from day 1 of study drug (including investigational agents, chemotherapy, and antibody-based therapy).
2. Patients currently receiving extracranial palliative radiation within 2 weeks from day 1 of study drug.
3. Patients who:

   1. Have had a major surgery or significant traumatic injury within 4 weeks from day 1 of study drug,
   2. Have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or
   3. Are anticipated to require major surgery during the course of the study.
4. Intolerance to PD-1/PD-L1 axis drug(s), or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including prior therapy with anti-tumor vaccines or other immune-stimulatory anti-tumor agents. (Intolerance: Toxicity that warrant no subsequent/further PD-1/PD-L1 therapy).
5. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent with the following exceptions:

   1. Intermittent steroids (not to exceed prednisone 10 mg every day or equivalent dosing) may be used on an as-needed basis (e.g., treatment for chemotherapy- related nausea, anorexia and fatigue.)
   2. Patients on physiologic replacement doses of steroids due to adrenal insufficiency for any reason may remain on these medications.
   3. Topical, inhaled or intra-articular corticosteroids
6. Symptomatic brain or leptomeningeal metastases, including patients who continue to require glucocorticoids and/or antiseizure therapy for brain or leptomeningeal metastases.

   1. Treated, asymptomatic metastases are permitted provided the patient has completed radiation at least 2 weeks prior to day 1 and has been off steroids for at least 2 weeks prior to day 1 of study drug.
   2. Stable (MRI or CT with contrast performed >4 weeks apart), untreated brain metastases are permitted if patient does not require steroids and/or antiseizure therapy is not required.
7. Presence of poorly controlled atrial fibrillation (ventricular heart rate >100 bpm) by EKG.
8. Previous history of CVA, TIA, angina pectoris, acute MI or history of recent re-perfusion procedures (e.g., PTCA), pulmonary embolus or untreated deep vein thrombosis within 6 months from day 1 of study drug. NOTE: Subjects with recent deep vein thrombosis and/or pulmonary embolus who have been therapeutically anti-coagulated for at least 6 weeks are eligible.
9. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study. Examples include but are not limited to:

   1. Active (acute or chronic) infections requiring treatment with antibiotics.
   2. Liver disease such as cirrhosis, chronic active or persistent hepatitis B or C or HIV.
   3. Age related macular degeneration, atypical hemolytic uremia syndrome, glomerulonephritis, or known autoimmune diseases.
   4. A concurrent diagnosis of a separate malignancy is allowed if clinically stable and does not require tumor-directed therapy
10. History of interstitial pneumonitis of autoimmune etiology (including immune checkpoint pneumonitis) which has been symptomatic and/or required treatment. History of radiation pneumonitis is allowed if the patient has recovered and does not currently require steroid therapy.
11. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to day 1 of study drug
12. Known autoimmune conditions requiring systemic immune suppressive therapy other than prednisone less than or equal to 10 mg.
13. Known history of HIV seropositivity or known acquired immunodeficiency syndrome (AIDS).
14. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. See Section 6.3.1.1 for a complete list of medically acceptable birth control methods.
15. Corrected QTc interval > 480 msec. If QTc interval is > 480 msec, then 2 additional ECGs should be obtained over a brief period (e.g., within 15-20 minutes) to confirm the abnormality. The average QTc interval will be determined from the 3 ECG tracings by manual evaluation and will be used to determine if the subject will be excluded from the study. The same method of QTc determination must be used throughout the subject's participation in the trial.
16. Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD), if any | 2 years
  The number and proportion of subjects at each dose level who experience a DLT
Time for the concentration of GT103 to reach half of the level administered | 2 years
Recommended phase II dose (RP2D) of GT103 | 2 years
  Recommended dose for the Phase II portion of the study

SECONDARY OUTCOMES:
Response Rate | 2 years
  Response rate is defined as the proportion of treated subjects with a complete or partial response. The response rate associated with the dose chosen to be the RP2D will also be estimated.
Progression-Free Survival | 2 years
  PFS is defined as the time between initiation of treatment and initial failure (disease progression or death). If the patient remains alive without disease progression at the time of analysis, PFS will be censored at the time of last follow-up. If the patient starts alternative anti-cancer therapy before progression, PFS will be censored at the time that the alternative treatment is initiated.
Overall Survival | 2 years
  OS is defined as the time between initiation of treatment and death.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Clarke, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Advent Health, Celebration, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clarke JM, Simon GR, Mamdani H, Gu L, Herndon JE 2nd, Stinchcombe TE, Ready N, Crawford J, Sonpavde G, Balevic S, Nixon AB, Campa M, Gottlin EB, Li H, Saxena R, He YW, Antonia S, Patz EF Jr. Complement factor H targeting antibody GT103 in refractory non-small cell lung cancer: a phase 1b dose escalation trial. Nat Commun. 2025 Jan 2;16(1):93. doi: 10.1038/s41467-024-55092-2. PMID 39747856